CLINICAL TRIAL: NCT00413751
Title: Effect of Brimonidine Tartrate Ophthalmic Solution 0.15% on Pupil Diameter in Normal Eyes
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: WRAMC WU #03-23004
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2006-12

CONDITIONS: Healthy
Keywords: Large pupils rendering night vision difficulties such as haloes, glare, and monocular diplopia
MeSH Terms: conditions — Diplopia | interventions — Brimonidine Tartrate

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Brimonidine tartrate ophthalmic solution 0.15% (Alphagan P)

SUMMARY:
The objective of this study is to evaluate the effect of brimonidine tartrate ophthalmic solution 0.15% (Alphagan P) on pupil diameter under different luminance conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult active duty personnel between 18 and 50 years of age with best corrected visual acuity of 20/20 or better.

Exclusion Criteria:

* Patients not meeting above stated age criteria
* Females that are pregnant or lactating (non pregnant females of childbearing potential will have pregnancy test prior to participating in study)
* History of serious ocular, neurological, cardiovascular disease
* History of severe systemic disease
* History of arrhythmias or high blood pressure
* Patients currently taking any type of ocular or systemic medications except multivitamins.
* Patients with abnormal pupil shape, Addie's pupil, anisocoria, or abnormal pupil defect.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Overall Officials: KRAIG S. BOWER, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States